CLINICAL TRIAL: NCT04897282
Title: Prospective Multicenter Trial to Determine the Efficacy and Outcome of the UCRI In-vitro Diagnostics Device to Detect Treatment Response Measured by Endoscopic Healing in Moderate to Severe Ulcerative Colitis Patients Treated With Anti-TNF-a.
Brief Title: Prospective Multicenter Trial to Determine the Efficacy and Outcome of the UCRI Biomarker Panel and Algorithm to Detect Mucosal Healing in Moderate to Severe Ulcerative Colitis Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glycominds, LLC (Industry)
Collaborators: University of California, Davis (Other); University of California, Irvine (Other); University of Chicago (Other); Weill Medical College of Cornell University (Other); Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UCRI-1020
Record Dates: First submitted 2021-04-26; First posted 2021-05-21 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, Serum, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: UCRI — Biomarker panel and algorithm

SUMMARY:
The purpose of this research study is to determine the efficacy and outcome of the UCRI (an in-vitro diagnostics device in the form of a blood test and an algorithm) as a tool to detect mucosal healing (level of inflammation in the colon) in people with moderate-to-severe ulcerative colitis treated with anti-TNFα. Another reason is to explore additional biomarkers in blood, stool or voice to detect disease activity and/or mucosal healing. A tool to detect the level of inflammation in the colon based on blood, stool or voice biomarkers may reduce the need or the number of invasive endoscopic procedures. This is an observational study and no treatment decision nor clinical intervention will be done based on results during this study and all collected data will be used only for the goal of the study and for obtaining FDA IDE for a follow-up study.

DETAILED DESCRIPTION:
At the early stage of mucosal inflammation in patients with inflammatory Bowel Diseases (IBD), neutrophils flood into intestinal mucosa, phagocytose pathogenic microbes, and promote mucosal healing and resolution of inflammation. However, large numbers of neutrophils infiltrating in the inflamed mucosa and accumulating in the epithelium cause damage of mucosal architecture, compromised epithelial barrier and production of inflammatory mediators. Novel neutrophil-related serum markers are emerging in the literature and are valid candidates to surrogate markers for mucosal healing (MH). NGAL is an anti-bacterial protein, whereas MMP-9 is a protein with enzymatic activity towards extracellular matrix (ECM) and non-ECM components, and is involved in cell signaling.

By formation of a complex between NGAL and MMP-9, NGAL is thought to protect MMP-9 from autodegradation. Cathelicidin LL37 is the 37 amino acids C-terminal part of human cationic antimicrobial protein (hCAP)18 and acts as an antimicrobial protein (AMP). It is found in lysosomes of macrophages and polymorphonuclear leukocytes (PMNs) as well as keratinocytes and plays a role in the early host response against invading pathogens via its broad-spectrum anti-microbial activity. The expression of LL37 was found to be increased in the inflamed mucosa of patients with UC and CD3. Moreover, increased colonic LL37 expression in macrophages and epithelium was observed during colitis in UC patients. Chitinase 3 like 1 (CHI3L1), also known as YKL-40, is a 39 kDa secreted glycoprotein member of the glycosyl hydrolase 18 family although it does not show chitotriosidase activity. It is secreted by macrophages and neutrophils and acts as a growth factor for vascular endothelial cells and fibroblasts.

In previous retrospective single-site study, consisting of serum samples and endoscopic evaluation before and after anti-TNFa treatment from 176 moderate-to-severe UC patients and 75 healthy controls, showed that the combined use of these markers is statistically significant and can accurately correlate with the Mayo endoscopic subscore (MES) and identify endoscopic response to infliximab (IFX) and adalimumab (ADM. An algorithm, the Ulcerative Colitis Response Index (UCRI), a unit-less index ranging from 0 (likely a responder) to 10 (likely a non-responder) was constructed and identified accentually the anti-TNFa non-responders' patients as measured by endoscopic assessment MES ≥2.

Glycominds, LLC (the "Sponsor") in support of the Crohn's and Colitis Foundation (CCF) IBD Venture will conduct this prospective multicenter longitudinal study in the U.S. Following screening and patient enrollment based on the inclusion and exclusion criteria Imaging, blood (serum) and fecal samples will be collected at certain predefined time points from bio naïve (naïve) and from anti-TNFa previously exposed (exposed) active (MES >2) UC patients that will start an anti-TNFa treatment or switch from one anti-TNFa type to another (infliximab-IFX or biosimilars, adalimumab-ADM, golimumab-GOM) at time of recruitment. Collected blood and stool samples will be used to determine the accuracy and prediction value of the UCRI biomarker panel and algorithm in comparison with endoscopic healing (measured as end point of MES ≤ 2) and in comparison to fecal Calprotectin. The IFX/ADM/GOM treatment decision and endoscopic evaluations before and after treatment initiation/switching will be done according to current clinical practice and Sponsor will not have any influence or responsibilities on those decisions.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis patients with Mayo Endoscopic Subscore of 2-3
* Start/switch anti -TNFa treatment
* Capable of at-home fCal testing

Exclusion Criteria:

* Pregnant women
* anti -TNFa dose escalation/adjustment
* Inability to undergo endoscopic assessments due to Proctitis
* Diagnosed with infectious diseases
* Steroid refractory

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be between the ages of 18 and 65 with a diagnosis of UC and MES = 2 or 3. and intend to start or switch anti-TNFa treatment. Women who are pregnant will also be excluded. Patients who are unable to undergo endoscopic evaluations due to proctitis will also be excluded, as well as patients who have a demonstrated history of steroid refraction. To avoid the 2nd endoscopic assessment time fluctuations patients under anti-TNFa dose escalation or dose adjustment regimen will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
UCRI panel validation | 24 weeks
  Accuracy as measured by ROC curve (receiver operating characteristic curve)
UCRI panel validation | 24 weeks
  PPV - Positive Predicative Value: proportions of positive tests that are true positive.
UCRI panel validation | 24 weeks
  NPV - Negative Predicative Value: proportions of negative tests that are true negative.

SECONDARY OUTCOMES:
fCal comparison analysis | 24 weeks
  As a secondary outcome a comparison analysis with fecal Calprotectin (fCal) at 250 ug/g cut-off value will be performed

OTHER OUTCOMES:
UCRI prediction value | 0-14 weeks
  The UCRI prediction value as survival analysis (longrank tests) of MES following anti-TNFa treatment. Event will be defined as MES<2

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Inflammatory Bowel Disease Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
MES, Treatment, MES, blinded patient characteristics and UCRI and fCal lab results will be shared with researchers.

REFERENCES:
- [Background] de Bruyn M, Ringold R, Martens E, Ferrante M, Van Assche G, Opdenakker G, Dukler A, Vermeire S. The Ulcerative Colitis Response Index for Detection of Mucosal Healing in Patients Treated With Anti-tumour Necrosis Factor. J Crohns Colitis. 2020 Feb 10;14(2):176-184. doi: 10.1093/ecco-jcc/jjz125. PMID 31628842
- [Background] Koon HW, Shih DQ, Chen J, Bakirtzi K, Hing TC, Law I, Ho S, Ichikawa R, Zhao D, Xu H, Gallo R, Dempsey P, Cheng G, Targan SR, Pothoulakis C. Cathelicidin signaling via the Toll-like receptor protects against colitis in mice. Gastroenterology. 2011 Nov;141(5):1852-63.e1-3. doi: 10.1053/j.gastro.2011.06.079. Epub 2011 Jul 14. PMID 21762664